CLINICAL TRIAL: NCT01583387
Title: Proof of Concept of the Effect of Water Intake on the DNA Adducts Formation
Brief Title: Effect of Water Intake on the DNA Adducts Formation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NU340
Record Dates: First submitted 2012-04-20; First posted 2012-04-24 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Healthy Adults
Keywords: healthy adults; urinary adducts; water intake

ARMS (2):
- 1= Intervention (Other)
  Interventions: Other: 1-Increased water intake regimen
- 2= Control (Other)
  Interventions: Other: 2-Non-modified water intake regimen

INTERVENTIONS:
Other: 1-Increased water intake regimen — Arm 1-Intervention
  Arms: 1= Intervention
Other: 2-Non-modified water intake regimen — Arm 2-Control
  Arms: 2= Control

SUMMARY:
The main purpose of the study is to assess the effect of water intake on the formation of 4-ABP DNA adducts.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects 20 to 45 years old (bound included)
* Smoker with at least 15 cigarettes/day
* Subjects with body mass index between 18 and 27kg/m2 (bound included)
* Subjects with a 3-meal diet (breakfast, lunch, dinner)
* Subjects who have an easy daily access to internet
* Subjects able to communicate well with the investigator and willing to comply the requirement of the study
* Subjects who have signed the form of informed consent and are registered to the French national welfare system

Exclusion Criteria:

* Subjects presenting evidence or history of severe or acute disease which could affect the results of the study or the vital status
* Subject practising physical activity in an intensive way according to the investigator judgment.
* Subject with a history of metabolic disease or with acute or chronic gastrointestinal disease except appendicectomy
* Subjects with diagnosed urinary tract disease
* Subjects with diagnosed lung or respiratory disease
* Subjects consuming regularly more than 3 units of alcohol per day
* Subjects who take drugs or presenting drug addiction (cannabis, opioids, amphetamines.)
* Subjects presenting a situation interfering with the outcomes of the study according to the investigator opinion
* Subjects working with painting, dry cleaning, dyes, pesticides, aluminium or alphalt
* Subjects who eat charcoaled food more than three meals/week
* Subjects with a vegetarian diet
* Subjects under local or general treatment which can modify measurements performed in the study, in particular the assessment of the hydration status (diuretic intake, or treatment interfering with metabolism and nutrition behaviour)
* Subjects planning to stop or reducing smoking or change their cigarette brand within the next 3 months
* Subjects in a situation which in the investigator's opinion could interfere with optimal participation in the present study or could constitute a special risk for the subject
* Subjects currently in a exclusion period following participation in another clinical trial
* Subjects having received 4500 euros indemnities for participation in clinical trials in the 12 previous months (including participation in the present study)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2011-02; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre CAP, Montpellier, France